CLINICAL TRIAL: NCT05828511
Title: Phase 1/2 Study of Linvoseltamab (Anti-BCMA X Anti-CD3 Bispecific Antibody) in Previously Untreated Patients With Symptomatic Multiple Myeloma
Brief Title: A Window of Opportunity Trial to Learn if Linvoseltamab is Safe and Well Tolerated, and How Well it Works in Adult Participants With Recently Diagnosed Multiple Myeloma Who Have Not Already Received Treatment
Acronym: LINKER-MM4
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5458-ONC-2158; 2022-500800-24-00 (EU CTIS Number)
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Newly Diagnosed Multiple Myeloma (NDMM); Autologous Stem Cell Transplantation (ASCT); Cluster of Differentiation 3 (CD3); BCMA; High Dose chemoTherapy (HDT); International Myeloma Working Group (IMWG)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Note: Phase 1 part B will be randomized 1:1. All other participants will be non-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 cohorts (Experimental): Linvoseltamab dose escalation (part A), dose expansion (part B), and evaluation of alternative step-up regimen (part C) for participants with NDMM who are treatment-naïve.
  Interventions: Drug: Linvoseltamab
- Phase 2 - transplant ineligible cohort (Experimental): Transplant-ineligible participants, enrolled in dose expansion, will receive selected linvoseltamab regimen until disease progression as per protocol.
  Interventions: Drug: Linvoseltamab
- Phase 2 - transplant eligible cohort (Experimental): Transplant-eligible participants, enrolled in dose expansion, will receive selected linvoseltamab regimen for a fixed duration of treatment as per protocol
  Interventions: Drug: Linvoseltamab

INTERVENTIONS:
Drug: Linvoseltamab — Linvoseltamab will be administered by intravenous (IV) infusion
  Other Names: REGN5458; Lynozyfic™

SUMMARY:
This study is researching an experimental drug called linvoseltamab (called "study drug"). The study is focused on participants with newly diagnosed multiple myeloma (NDMM) who are eligible for high dose chemotherapy with autologous stem cell transplantation (transplant-eligible) or ineligible for autologous stem cell transplantation (transplant-ineligible).

The aim of this clinical trial is to study the safety, tolerability (how the body reacts to the drug), and effectiveness (tumor shrinkage) of linvoseltamab in study participants with NDMM as a first step in determining if the study drug has a role in the treatment of NDMM.

This study consists of 2 phases:

* In Phase 1 Parts A and B, the study drug will be given to participants to study the side effects of the study drug and to establish the regimen (initial doses and full dose) of the study drug to be given to participants in Phase 2.
* In Phase 1 Part C, the study drug will be given to participants to study the side effects when using different initial doses of the study drug.
* In Phase 2, the study drug will be given to more participants to continue to assess the side effects of the study drug and to evaluate the activity of the study drug to shrink the tumor (multiple myeloma) in participants with NDMM.

The study is looking at several research questions, including:

* What side effects may happen from taking linvoseltamab?
* What the right dosing regimen is for linvoseltamab?
* How many participants treated with linvoseltamab have improvement of their disease and for how long?
* The effects of linvoseltamab study treatment before and after transplant
* How much linvoseltamab is in the blood at different times?
* Whether the body makes antibodies against linvoseltamab (which could make the drug less effective or could lead to side effects).

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
2. Confirmed diagnosis of symptomatic Multiple Myeloma (MM) by International Myeloma Working Group (IMWG) diagnosis criteria, as described in the protocol
3. Response-evaluable myeloma, according to the 2016 IMWG response criteria, as defined in the protocol
4. No prior therapy for MM, with the exception of prior emergent or palliative radiation and up to 1 month of single-agent corticosteroids, with washout periods as per the protocol
5. Participants must have evidence of adequate bone marrow reserves and hepatic, renal and cardiac function as defined in the protocol
6. Participants must be age <70 and have adequate hepatic, renal, pulmonary and cardiac function to be considered transplant-eligible. The specific thresholds for adequate organ function are as per institutional guidance.

Key Exclusion Criteria:

1. Receiving any concurrent investigational agent with known or suspected activity against MM, or agents targeting the A proliferation-inducing ligand (APRIL)/ Transmembrane activator and calcium modulator and cyclophilin ligand interactor (TACI)/BCMA axis
2. Known Central Nervous System (CNS) involvement with MM, known or suspected Progressive Multifocal Leukoencephalopathy (PML), a history of neurocognitive conditions, or CNS movement disorder, or history of seizure within 12 months prior to study enrollment
3. Rapidly progressive symptomatic disease, (e.g. progressing renal failure or hypercalcemia not responsive to standard medical interventions), in urgent need of treatment with chemotherapy
4. Diagnosis of non-secretory MM, active plasma cell leukemia primary light-chain (AL) amyloidosis, Waldenström macroglobulinemia (lymphoplasmacytic lymphoma), or known POEMS syndrome (Plasma cell dyscrasia with polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, and Skin changes)

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2035-11-02 (Estimated); Study Completion 2035-11-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | End of the Observation period; up to day 28
  Phase 1
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 1
Severity of TEAEs | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 1
Incidence of Adverse Events of Special Interest (AESIs) | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 1
Severity of AESIs | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 1
Proportion of participants with a Very Good Partial Response (VGPR) or better using the International Myeloma Working Group (IMWG) response criteria | Up to 5 years
  Phase 2
Proportion of participants achieving Minimal Residual Disease (MRD) negative status (at 10^-5) after induction with consolidation therapy | Up to 5 years
  Phase 2 Transplant-eligible cohort
Proportion of participants achieving MRD-negative status (at 10^-5) after induction without consolidation therapy | Up to 5 years
  Phase 2 Transplant-eligible cohort
Proportion of participants achieving MRD-negative status as their best response after treatment period I with continuing to treatment period II | Up to 5 years
  Phase 2 Transplant-ineligible cohort
Proportion of participants achieving MRD-negative status as their best response after treatment period I without continuing to treatment period II | Up to 5 years
  Phase 2 Transplant ineligible cohort

SECONDARY OUTCOMES:
Concentrations of Linvoseltamab in serum | Post-Last Linvoseltamab Dose, up to 12 weeks
  Phases 1 and 2
Concentrations of total soluble B-Cell Maturation Antigen (BCMA) | Post-Last Linvoseltamab Dose, up to 12 weeks
  Phases 1 and 2
Incidence of Anti-Drug Antibodies (ADAs) to Linvoseltamab | Post-Last Linvoseltamab Dose, up to 30 days
  Phases 1 and 2
Magnitude of ADAs to Linvoseltamab | Post-Last Linvoseltamab Dose, up to 30 days
  Phases 1 and 2
Objective Response Rate (ORR) measured using the IMWG criteria | Up to 5 years
  Phase 1
Duration Of Response (DOR) measured using the IMWG criteria | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 1
Progression-Free Survival (PFS) measured using the IMWG criteria | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 1
Proportion of participants achieving MRD-negative status (at 10^-5) in participants with NDMM measured using the IMWG criteria | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 1
Incidence of TEAEs | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
Severity of TEAEs | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
Incidence of AESIs | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
Severity of AESIs | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
ORR of participants deemed transplant-eligible and transplant-ineligible by the treating physician | Up to 5 years
  Phase 2
MRD-negative status of participants deemed transplant-eligible and transplant-ineligible by the treating physician | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
DOR of participants deemed transplant-eligible and transplant-ineligible by the treating physician | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
PFS of participants deemed transplant-eligible and transplant-ineligible by the treating physician | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
Overall Survival (OS) of participants deemed transplant-eligible and transplant-ineligible by the treating physician | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
Time To Response (TTR) as measured using the IMWG criteria | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
ORR by risk levels | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
MRD-negative status by risk levels | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
DOR by risk levels | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
TTR by risk levels | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
PFS by risk levels | Post-Last Linvoseltamab Dose, up to 90 days
  Phase 2
Incidence of MRD-negative status | Up to 5 years
  Phase 2
Cluster of Differentiation 34+ (CD34+) stem cell yield | At cycle 4 of induction (each cycle is 28 days long)
  Phase 2 Transplant-eligible cohort
Time to neutrophil engraftment | Up to 100 days post-transplant
  Phase 2 Transplant-eligible cohort
Time to platelet engraftment | Up to 100 days post-transplant
  Phase 2 Transplant-eligible cohort
PFS after ASCT followed by 3 cycles of linvoseltamab | Up to 5 years
  Phase 2 Transplant-eligible cohort

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (32):
- United States (13):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - UC Irvine Health, Orange, California
  - Colorado Blood Cancer Institute/SCRI, Denver, Colorado
  - Norton Cancer Institute, Louisville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Perlmutter Cancer Center, New York, New York
  - Columbia University _ New York Presbyterian, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Health System (DUHS), Durham, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- France (8):
  - Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers, Nouvelle-Aquitaine
  - CHU De Lille, Lille
  - Centre Hospitalier Universitaire (CHU) Montpellier, Montpellier
  - Hopital Saint Louis, Paris
  - Hopital Pitié Salpetriere APHP, Paris
  - Hopital Prive d'Antony, Antony, Île-de-France Region
  - Hopital Necker, Paris, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region
- Spain (11):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Quiron Salud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario Doctor Balmis Alicante, Alicante, Valencia
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala dOncologia (ICO Hospitalet), Barcelona
  - Universitary Hospital La Princesa, Madrid
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - La Fe University Hospital, Valencia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/